## **COVER PAGE**

**Study title:** Simultaneous tDCS and Computerised Gamified Short-term Memory Task Feasibility (ACTTDCS-FG)

NCT ID: Not yet assigned

**Document type:** Consent form

**Original date of the document:** September 5, 2021

## Consent form for participation in a health research project

Study title: "Pre-symptomatic Alzheimer's disease: Cognitive training and transcranial direct current stimulation (tDCS)"

## **Declaration from the participant:**

Nama

I hereby consent to participate in the study, "Pre-symptomatic Alzheimer's disease: Cognitive training and transcranial direct current stimulation (tDCS)", for which I will complete a cognitive task on a tablet in combination with headset-delivered transcranial direct current stimulation (tDCS) on three different occasions.

I declare that I have received sufficient written and oral information about the study to be able to consent to participate herein. I know it's voluntary to participate and that I can withdraw from the study at any time without having to give a reason and without any consequences for any current or future treatment I may require.

I have been informed that I can get a copy of the signed consent form, if I desire.

| Name: | |
|---|---|
| Date: | Signature: |
| <b>Declaration from the</b> | member of scientific staff giving the information: |
| to ask questions about of<br>wishes to participate he<br>the right to withdraw fr | e participant has received written and oral information about the study, has had time each part of the study and has been given sufficient time to consider if he or she trein. The participant has been thoroughly informed about his or her rights, including om the study at any time without needing to give a reason and without it having any arrent or future treatments they may require. |
| Date: | Signature: |